CLINICAL TRIAL: NCT02062008
Title: Validation of Combined PET-MR Quantitative Parameters for Cardiac Applications
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding to continue.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Combined PET-MRI
Record Dates: First submitted 2014-02-07; First posted 2014-02-13 (Estimated); Results first posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-05

CONDITIONS: Cardiac Disease
Keywords: Positron Emission Tomography-Magnetic Resonance Imaging; Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiac patients receiving PET/MR (Other): PET-MRI with intravenous Gadolinium and FDG. The entire study will take approximately one hour.
  Interventions: Device: PET-MRI

INTERVENTIONS:
Device: PET-MRI — PET-MRI with intravenous Gadolinium and FDG. The entire study will take approximately one hour.

SUMMARY:
The purpose of this study is to understand how simultaneous PET/MR acquisition can provide novel qualitative and quantitative biomarkers to guide clinical intervention and predict prognosis of patients with cardiovascular disease.

DETAILED DESCRIPTION:
* To compare regional myocardial uptake of FDG on images obtained on a standard PET camera with the new PET/MR camera, in patients with coronary artery disease.
* To compare viability maps obtained with cardiac MR images and FDG-PET for delineation of myocardial infarct core and border zone, in patients with coronary artery disease.
* To correlate MRI myocardial strain with relative myocardial FDG uptake in patients with a previous myocardial infarction.
* To interrogate if simultaneous acquisition of cardiac PET and viability cardiac MR differ from acquisitions obtained independently, with special focus on attenuation correction methods
* To combined MRI scar map with FDG-PET uptake in patients with cardiac sarcoidosis and myocarditis.
* To correlate morphologic characteristics of atherosclerotic disease in the thoracic and abdominal aorta with FDG uptake and ferumoxytol enhancement, as a marker of inflammation.
* To evaluate cardiac strain and myocardial scar burden in obese patients with and without diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with ischemic and non-ischemic cardiac disease referred for cardiac PET for viability imaging.

Exclusion Criteria:

* Contraindications for MRI, including cardiac pacemaker, claustrophobia, retained metallic foreign body, cochlear implant, Aneurysm clip in the brain, pregnancy and eGFR less than 45%.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-02-10 (Actual); Study Completion 2018-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen G Ordovas, MD,MAS, Principal Investigator — Assistent Professor
Locations (1):
- UCSF University of California in San Francisco, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cardiac Patients Receiving PET/MR
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cardiac Patients Receiving PET/MR
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Quality PET and PET/MR Images With Regional Myocardial Uptake of 18F-Fluorodeoxyglucose (FDG) in Participants Without Overt Diagnosis of Ischemic Coronary Artery Disease.
Description: Visual analysis of collected image pairs. Evaluated by experienced imaging providers as yes or no.
Time Frame: 2 hours
Measure: Number; unit: quality image
Arm/Group | Cardiac Patients Receiving PET/MR
Number analyzed (Participants) | 2
quality image | 2

ADVERSE EVENTS:
Time Frame: One year
Description: Imaging agent FDG has demonstrated a minimal risk, with no allergy or other local or systemic side effects.
Arm/Group | Cardiac Patients Receiving PET/MR
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT02062008/Prot_SAP_000.pdf